CLINICAL TRIAL: NCT04973085
Title: Effect of a Novel Cooling Device on Brain Temperature
Brief Title: Neck Cooling as a Non-Invasive Method to Lower Brain Temperature in Healthy Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Vermont (Other)
Collaborators: Becton, Dickinson and Company (Industry)
Responsible Party: Principal Investigator, Adam Sprouse Blum, Assistant Professor of Neurological Sciences, University of Vermont
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: STUDY00001312
Record Dates: First submitted 2021-06-28; First posted 2021-07-22 (Actual); Results first posted 2023-09-13 (Actual); Last update posted 2023-09-13 (Actual); Status verified 2023-08

CONDITIONS: Healthy
Keywords: targeted temperature management; brain temperature; brain cooling; neck cooling

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Cold circulated water (Experimental): Cold water circulated through an adhesive wrap applied to the front of the neck.
  Interventions: Device: Cold circulated water
- Body-temperature circulated water (Active Comparator): Body-temperature water circulated through an adhesive wrap applied to the front of the neck.
  Interventions: Device: Body-temperature circulated water

INTERVENTIONS:
Device: Cold circulated water — Cold water was circulated through an adhesive wrap applied to the front of the neck, overlying the carotid arteries, for 120 minutes. MR thermometry was used to measure core brain temperature in 1-minute intervals throughout the intervention. On a different day, subjects crossed over and repeated the intervention in the other study arm (i.e., cold went to body-temperature, and vice-versa).
  Arms: Cold circulated water
Device: Body-temperature circulated water — Body-temperature water was circulated through an adhesive wrap applied to the front of the neck, overlying the carotid arteries, for 120 minutes. MR thermometry was used to measure core brain temperature in 1-minute intervals throughout the intervention. On a different day, subjects crossed over and repeated the intervention in the other study arm (i.e., cold went to body-temperature, and vice-versa).
  Arms: Body-temperature circulated water

SUMMARY:
The objective of this study was to clarify whether neck cooling can be used to non-invasively lower brain temperature in healthy adults.

DETAILED DESCRIPTION:
Healthy adults were randomized to undergo an intervention in which either cold or body-temperature water was circulated through an adhesive wrap applied to the front of their necks, overlying the carotid arteries, for 120 minutes. After their first intervention, subjects crossed over (i.e., cold went to body-temperature, and vice-versa) on a separate day. Brain temperature was measured in one-minute intervals using MR thermometry.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults aged 18-65 years

Exclusion Criteria:

* Pregnancy
* Contraindications to MRI (e.g. claustrophobia, metallic implants, etc.)
* Signs of ulcerations, burns, hives or rash where the neck wrap is applied
* History of Raynaud's disease, venous or arterial occlusive disease (e.g. carotid stenosis), cryoprecipitation disorders (e.g. cryoglobulinemia) and pernio (also known as chilblains)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2021-07-22 (Actual); Primary Completion 2022-03-03 (Actual); Study Completion 2022-03-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Adam S Sprouse Blum, MD, Principal Investigator — University of Vermont
Locations (1):
- University of Vermont & State Agricultural College, Burlington, Vermont, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wang H, Wang B, Normoyle KP, Jackson K, Spitler K, Sharrock MF, Miller CM, Best C, Llano D, Du R. Brain temperature and its fundamental properties: a review for clinical neuroscientists. Front Neurosci. 2014 Oct 8;8:307. doi: 10.3389/fnins.2014.00307. eCollection 2014. PMID 25339859
- [Background] Wass CT, Lanier WL, Hofer RE, Scheithauer BW, Andrews AG. Temperature changes of > or = 1 degree C alter functional neurologic outcome and histopathology in a canine model of complete cerebral ischemia. Anesthesiology. 1995 Aug;83(2):325-35. doi: 10.1097/00000542-199508000-00013. PMID 7631955
- [Background] Arrich J, Holzer M, Havel C, Mullner M, Herkner H. Hypothermia for neuroprotection in adults after cardiopulmonary resuscitation. Cochrane Database Syst Rev. 2016 Feb 15;2(2):CD004128. doi: 10.1002/14651858.CD004128.pub4. PMID 26878327
- [Background] Jiang JY, Xu W, Yang PF, Gao GY, Gao YG, Liang YM, Yin XL, Zhu C. Marked protection by selective cerebral profound hypothermia after complete cerebral ischemia in primates. J Neurotrauma. 2006 Dec;23(12):1847-56. doi: 10.1089/neu.2006.23.1847. PMID 17184193
- [Background] Natale JA, D'Alecy LG. Protection from cerebral ischemia by brain cooling without reduced lactate accumulation in dogs. Stroke. 1989 Jun;20(6):770-7. doi: 10.1161/01.str.20.6.770. PMID 2728044
- [Background] Noguchi Y, Nishio S, Kawauchi M, Asari S, Ohmoto T. A new method of inducing selective brain hypothermia with saline perfusion into the subdural space: effects on transient cerebral ischemia in cats. Acta Med Okayama. 2002 Dec;56(6):279-86. doi: 10.18926/AMO/31690. PMID 12685856
- [Background] Davidson JO, Wassink G, Yuill CA, Zhang FG, Bennet L, Gunn AJ. How long is too long for cerebral cooling after ischemia in fetal sheep? J Cereb Blood Flow Metab. 2015 May;35(5):751-8. doi: 10.1038/jcbfm.2014.259. Epub 2015 Jan 21. PMID 25605291
- [Background] Kuluz JW, Gregory GA, Yu AC, Chang Y. Selective brain cooling during and after prolonged global ischemia reduces cortical damage in rats. Stroke. 1992 Dec;23(12):1792-6; discussion 1797. doi: 10.1161/01.str.23.12.1792. PMID 1448830
- [Background] Dumitrascu OM, Lamb J, Lyden PD. Still cooling after all these years: Meta-analysis of pre-clinical trials of therapeutic hypothermia for acute ischemic stroke. J Cereb Blood Flow Metab. 2016 Jul;36(7):1157-64. doi: 10.1177/0271678X16645112. Epub 2016 Apr 18. PMID 27089911
- [Background] Torok E, Klopotowski M, Trabold R, Thal SC, Plesnila N, Scholler K. Mild hypothermia (33 degrees C) reduces intracranial hypertension and improves functional outcome after subarachnoid hemorrhage in rats. Neurosurgery. 2009 Aug;65(2):352-9; discussion 359. doi: 10.1227/01.NEU.0000345632.09882.FF. PMID 19625915
- [Background] Dietrich WD, Bramlett HM. Therapeutic hypothermia and targeted temperature management for traumatic brain injury: Experimental and clinical experience. Brain Circ. 2017 Oct-Dec;3(4):186-198. doi: 10.4103/bc.bc_28_17. Epub 2017 Dec 29. PMID 30276324
- [Background] Bennett AE, Hoesch RE, DeWitt LD, Afra P, Ansari SA. Therapeutic hypothermia for status epilepticus: A report, historical perspective, and review. Clin Neurol Neurosurg. 2014 Nov;126:103-9. doi: 10.1016/j.clineuro.2014.08.032. Epub 2014 Sep 4. PMID 25240131
- [Background] Schwab M, Bauer R, Zwiener U. Mild hypothermia prevents the occurrence of cytotoxic brain edema in rats. Acta Neurobiol Exp (Wars). 1998;58(1):29-35. doi: 10.55782/ane-1998-1256. PMID 9583185
- [Background] Geocadin RG, Wijdicks E, Armstrong MJ, Damian M, Mayer SA, Ornato JP, Rabinstein A, Suarez JI, Torbey MT, Dubinsky RM, Lazarou J. Practice guideline summary: Reducing brain injury following cardiopulmonary resuscitation: Report of the Guideline Development, Dissemination, and Implementation Subcommittee of the American Academy of Neurology. Neurology. 2017 May 30;88(22):2141-2149. doi: 10.1212/WNL.0000000000003966. Epub 2017 May 10. PMID 28490655
- [Background] Jacobs SE, Berg M, Hunt R, Tarnow-Mordi WO, Inder TE, Davis PG. Cooling for newborns with hypoxic ischaemic encephalopathy. Cochrane Database Syst Rev. 2013 Jan 31;2013(1):CD003311. doi: 10.1002/14651858.CD003311.pub3. PMID 23440789
- [Background] Crossley S, Reid J, McLatchie R, Hayton J, Clark C, MacDougall M, Andrews PJ. A systematic review of therapeutic hypothermia for adult patients following traumatic brain injury. Crit Care. 2014 Apr 17;18(2):R75. doi: 10.1186/cc13835. PMID 24742169
- [Background] Karnatovskaia LV, Wartenberg KE, Freeman WD. Therapeutic hypothermia for neuroprotection: history, mechanisms, risks, and clinical applications. Neurohospitalist. 2014 Jul;4(3):153-63. doi: 10.1177/1941874413519802. PMID 24982721
- [Background] Geurts M, Macleod MR, Kollmar R, Kremer PH, van der Worp HB. Therapeutic hypothermia and the risk of infection: a systematic review and meta-analysis. Crit Care Med. 2014 Feb;42(2):231-42. doi: 10.1097/CCM.0b013e3182a276e8. PMID 23989182
- [Background] Khera R, Humbert A, Leroux B, Nichol G, Kudenchuk P, Scales D, Baker A, Austin M, Newgard CD, Radecki R, Vilke GM, Sawyer KN, Sopko G, Idris AH, Wang H, Chan PS, Kurz MC. Hospital Variation in the Utilization and Implementation of Targeted Temperature Management in Out-of-Hospital Cardiac Arrest. Circ Cardiovasc Qual Outcomes. 2018 Nov;11(11):e004829. doi: 10.1161/CIRCOUTCOMES.118.004829. PMID 30571336
- [Background] Stanger D, Kawano T, Malhi N, Grunau B, Tallon J, Wong GC, Christenson J, Fordyce CB. Door-to-Targeted Temperature Management Initiation Time and Outcomes in Out-of-Hospital Cardiac Arrest: Insights From the Continuous Chest Compressions Trial. J Am Heart Assoc. 2019 May 7;8(9):e012001. doi: 10.1161/JAHA.119.012001. PMID 31055981
- [Background] Kurisu K, Yenari MA. Therapeutic hypothermia for ischemic stroke; pathophysiology and future promise. Neuropharmacology. 2018 May 15;134(Pt B):302-309. doi: 10.1016/j.neuropharm.2017.08.025. Epub 2017 Aug 19. PMID 28830757
- [Background] Ohta H, Terao Y, Shintani Y, Kiyota Y. Therapeutic time window of post-ischemic mild hypothermia and the gene expression associated with the neuroprotection in rat focal cerebral ischemia. Neurosci Res. 2007 Mar;57(3):424-33. doi: 10.1016/j.neures.2006.12.002. Epub 2007 Jan 8. PMID 17212971
- [Background] Thoresen M, Tooley J, Liu X, Jary S, Fleming P, Luyt K, Jain A, Cairns P, Harding D, Sabir H. Time is brain: starting therapeutic hypothermia within three hours after birth improves motor outcome in asphyxiated newborns. Neonatology. 2013;104(3):228-33. doi: 10.1159/000353948. Epub 2013 Sep 12. PMID 24030160
- [Background] Nybo L, Wanscher M, Secher NH. Influence of intranasal and carotid cooling on cerebral temperature balance and oxygenation. Front Physiol. 2014 Feb 27;5:79. doi: 10.3389/fphys.2014.00079. eCollection 2014. PMID 24578693
- [Background] Curran EJ, Wolfson DL, Watts R, Freeman K. Cold Blooded: Evaluating Brain Temperature by MRI During Surface Cooling of Human Subjects. Neurocrit Care. 2017 Oct;27(2):214-219. doi: 10.1007/s12028-017-0389-4. PMID 28352966
- [Background] Abou-Chebl A, Sung G, Barbut D, Torbey M. Local brain temperature reduction through intranasal cooling with the RhinoChill device: preliminary safety data in brain-injured patients. Stroke. 2011 Aug;42(8):2164-9. doi: 10.1161/STROKEAHA.110.613000. Epub 2011 Jun 16. PMID 21680904
- [Background] Vanderpol J, Bishop B, Matharu M, Glencorse M. Therapeutic effect of intranasal evaporative cooling in patients with migraine: a pilot study. J Headache Pain. 2015 Jan 26;16:5. doi: 10.1186/1129-2377-16-5. PMID 25623151
- [Background] Covaciu L, Weis J, Bengtsson C, Allers M, Lunderquist A, Ahlstrom H, Rubertsson S. Brain temperature in volunteers subjected to intranasal cooling. Intensive Care Med. 2011 Aug;37(8):1277-84. doi: 10.1007/s00134-011-2264-7. Epub 2011 Jun 7. PMID 21647717
- [Background] Poli S, Purrucker J, Priglinger M, Sykora M, Diedler J, Rupp A, Bulut C, Hacke W, Hametner C. Safety evaluation of nasopharyngeal cooling (RhinoChill(R)) in stroke patients: an observational study. Neurocrit Care. 2014 Feb;20(1):98-105. doi: 10.1007/s12028-013-9904-4. PMID 24026521
- [Background] Harris S, Bansbach J, Dietrich I, Kalbhenn J, Schmutz A. RhinoChill((R))-more than an "ice-cream headache (1)" serious adverse event related to transnasal evaporative cooling. Resuscitation. 2016 Jun;103:e5-e6. doi: 10.1016/j.resuscitation.2016.01.036. Epub 2016 Mar 12. No abstract available. PMID 26980347
- [Background] Gorbach AM, Heiss J, Kufta C, Sato S, Fedio P, Kammerer WA, Solomon J, Oldfield EH. Intraoperative infrared functional imaging of human brain. Ann Neurol. 2003 Sep;54(3):297-309. doi: 10.1002/ana.10646. PMID 12953262
- [Background] Keller E, Mudra R, Gugl C, Seule M, Mink S, Frohlich J. Theoretical evaluations of therapeutic systemic and local cerebral hypothermia. J Neurosci Methods. 2009 Apr 15;178(2):345-9. doi: 10.1016/j.jneumeth.2008.12.030. Epub 2009 Jan 9. PMID 19167429
- [Background] Krejza J, Arkuszewski M, Kasner SE, Weigele J, Ustymowicz A, Hurst RW, Cucchiara BL, Messe SR. Carotid artery diameter in men and women and the relation to body and neck size. Stroke. 2006 Apr;37(4):1103-5. doi: 10.1161/01.STR.0000206440.48756.f7. Epub 2006 Feb 23. PMID 16497983
- [Background] Hall, L. D., & Talagala, S. L. (1985). Mapping of pH and temperature distribution using chemical-shift-resolved tomography. Journal of Magnetic Resonance (1969), 65(3), 501-505.
- [Background] De Poorter J, De Wagter C, De Deene Y, Thomsen C, Stahlberg F, Achten E. Noninvasive MRI thermometry with the proton resonance frequency (PRF) method: in vivo results in human muscle. Magn Reson Med. 1995 Jan;33(1):74-81. doi: 10.1002/mrm.1910330111. PMID 7891538
- [Background] Ishihara Y, Calderon A, Watanabe H, Okamoto K, Suzuki Y, Kuroda K, Suzuki Y. A precise and fast temperature mapping using water proton chemical shift. Magn Reson Med. 1995 Dec;34(6):814-23. doi: 10.1002/mrm.1910340606. PMID 8598808
- [Background] Harris B, Andrews PJ, Murray GD, Forbes J, Moseley O. Systematic review of head cooling in adults after traumatic brain injury and stroke. Health Technol Assess. 2012;16(45):1-175. doi: 10.3310/hta16450. PMID 23171713

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 22 subjects were screened for study eligibility between July, 2021 and February, 2022.
Pre-assignment Details: Subjects were randomized to either the cold or body-temperature water arm at the MRI research center immediately prior to their first intervention.
Groups:
- Cold (Intervention 1) Then Body-temperature (Intervention 2) Circulated Water: Participants first underwent the intervention with cold circulated water. Then, on a separate day, they repeated the intervention with body-temperature water.
- Body-temperature (Intervention 1) Then Cold (Intervention 2) Circulated Water: Participants first underwent the intervention with body-temperature circulated water. Then, on a separate day, they repeated the intervention with cold water.
Period: First Intervention
Arm/Group | Cold (Intervention 1) Then Body-temperature (Intervention 2) Circulated Water | Body-temperature (Intervention 1) Then Cold (Intervention 2) Circulated Water
Started | 10 | 12
Completed | 9 | 12
Not Completed | 1 | 0
Not completed — Claustrophobia in the MRI machine. | 1 | 0
Period: Second Intervention
Arm/Group | Cold (Intervention 1) Then Body-temperature (Intervention 2) Circulated Water | Body-temperature (Intervention 1) Then Cold (Intervention 2) Circulated Water
Started | 9 | 12
MRI Adjusted Protocol (The data from the first 5 subjects was used to modify the MRI protocol to improve the accuracy of the results. All subjects who were scanned using the modified MRI protocol were analyzed.) | 7 | 9
Completed | 7 | 9
Not Completed | 2 | 3

BASELINE CHARACTERISTICS:
Groups:
- Analyzed Participants: All analyzed participants.
- Participants Used to Modify MRI Protocol: Participants whose data was used to modify the MRI protocol.
- Total: Total of all reporting groups
Arm/Group | Analyzed Participants | Participants Used to Modify MRI Protocol | Total
Number analyzed (Participants) | 17 | 5 | 22
Age, Continuous [Mean (Standard Deviation); unit: years] | 31.1 (10.9) | 21.1 (1.8) | 28.9 (10.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 2 | 12
  Male | 7 | 3 | 10
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Change in Brain Temperature
Description: During each intervention, core brain temperature was measured non-invasively, in one-minute increments, using MR thermometry. The change in brain temperature was calculated as the difference of differences between the cold and body-temperature interventions, after 1 hour.
Time Frame: 60 minutes
Population: Two participants were excluded from the analyses, including one who was not able to complete the interventions due to claustrophobia, and one who had incomplete data due to documented head movement.
Measure: Median (95% Confidence Interval); unit: degrees Celsius
Groups:
- Cold Circulated Water: Participants undergoing the intervention with cold circulated water.
- Body-temperature Circulated Water: Participants undergoing the intervention with body-temperature circulated water.
Arm/Group | Cold Circulated Water | Body-temperature Circulated Water
Number analyzed (Participants) | 15 | 15
degrees Celsius | -0.23 [-0.37 to -0.10] | -0.03 [-0.14 to 0.09]
Statistical Analysis 1: Comparison: Cold Circulated Water vs Body-temperature Circulated Water; Test type: Other; p = 0.02, t-test, 2 sided

2. Secondary Outcome: Modified Bedside Shivering Assessment
Time Frame: 120 minutes
Measure: Count of Participants; unit: Participants
Arm/Group | Cold Circulated Water | Body-temperature Circulated Water
Number analyzed (Participants) | 15 | 15
Participants
  Number of participants with BSAS score = 0 (none) | 15 | 15
  Number of participants with BSAS score = 1 (mild) | 0 | 0
  Number of participants with BSAS score = 2 (moderate) | 0 | 0
  Number of participants with BSAS score = 3 (severe) | 0 | 0

3. Secondary Outcome: Systolic Blood Pressure
Description: Change in systolic blood pressure during the intervention.
Time Frame: 120 minutes
Measure: Median (95% Confidence Interval); unit: mmHg
Arm/Group | Cold Circulated Water | Body-temperature Circulated Water
Number analyzed (Participants) | 15 | 15
mmHg | -1.7 [-4.8 to 1.4] | 2.9 [0.4 to 5.5]

4. Secondary Outcome: Diastolic Blood Pressure
Time Frame: 120 minutes
Measure: Median (95% Confidence Interval); unit: mmHg
Arm/Group | Cold Circulated Water | Body-temperature Circulated Water
Number analyzed (Participants) | 15 | 15
mmHg | 2.8 [0.5 to 5.1] | 0.8 [-1.7 to 3.3]

5. Secondary Outcome: Heart Rate
Time Frame: 120 minutes
Measure: Median (95% Confidence Interval); unit: beats per minute
Arm/Group | Cold Circulated Water | Body-temperature Circulated Water
Number analyzed (Participants) | 15 | 15
beats per minute | -2.0 [-4.0 to 0.1] | 0.2 [-2.8 to 3.3]

ADVERSE EVENTS:
Time Frame: 120 minutes
Description: Adverse event information was collected immediately after each intervention, by asking participants: "Did you experience any adverse effects during the intervention? If yes, please explain."
Groups:
- Cold Circulated Water: Adverse events occurring during the cold intervention.
- Body-temperature Circulated Water: Adverse events occurring during the body-temperature intervention.
Arm/Group | Cold Circulated Water | Body-temperature Circulated Water
All-Cause Mortality (participants affected / at risk) | 0/22 | 0/21
Serious Adverse Events (participants affected / at risk) | 0/22 | 0/21
Other Adverse Events (participants affected / at risk) | 5/22 | 2/21
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cold Circulated Water (N=22) | Body-temperature Circulated Water (N=21)
Claustrophobia in the MRI scanner (Investigations) | 1 (1) | 0 (0)
Skin discomfort (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Stiff neck (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 1 (1)
Dizziness (Ear and labyrinth disorders) | 1 (1) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-09-29): https://cdn.clinicaltrials.gov/large-docs/85/NCT04973085/Prot_SAP_000.pdf